CLINICAL TRIAL: NCT05579340
Title: Post-Operative Exercise Training in Patients With Metastatic Colorectal Cancer
Brief Title: Postoperative Exercise Training and Colorectal Cancer Liver Metastasis
Acronym: mCRC-POET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christina Yfanti, Postdoctoral researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: mCRC-POET
Record Dates: First submitted 2022-09-22; First posted 2022-10-13 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Cancer Metastatic to Liver; Cancer Colorectal
MeSH Terms: conditions — Colonic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention)
- Ex1 (Experimental): Low exercise volume (150 min/week)
  Interventions: Other: Exercise
- Ex2 (Experimental): High exercise volume (300 min/week)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 6 months of combined aerobic and resistance exercise
  Arms: Ex1; Ex2

SUMMARY:
Up to 25% of colorectal cancer (CRC) patients are diagnosed with liver metastases, which is the most common site of metastasis, already during the primary tumor diagnosis. Another 30% of the patients will develop liver metastases at a later stage. Even though patient can be treated by surgical resection of the metastatic tumor, 50-75% of the patients experience a relapse in less than two years. Due to the high probability of relapse, mCRC patients undergo multiple rounds of surgery and adjuvant treatment (chemotherapy/radiotherapy) which results in substantial physical de-conditioning.

Physical activity has been shown to increase the progression-free survival rates in mCRC patients, when applied post-diagnosis. Increased cardiorespiratory fitness (VO2peak) at the time of diagnosis among CRC individuals has been associated with lower risk of all-cause mortality. Although data on the effect of chronic exercise on VO2peak have emerged, thus far, there is no randomized clinical trial that has investigated the effects of exercise training in mCRC patients early after surgical treatment with curative intent.

Therefore, this project aims to address the beneficial effect of structured exercise training primarily on VO2peak and tumor recurrence in mCRC patients immediately after surgical treatment and while they are undergoing adjuvant chemotherapy/radiotherapy.

A total of 66 participants will be recruited from the Department of Surgery and Transplantation, Rigshospitalet and randomly allocated to a standard care control group (n=22), standard care plus 150 min/week exercise training (n=22) or standard care plus 300 min/week exercise training (n=22). Participants will undergo exercise training for 6 months, starting immediately after surgery, and they will be followed for additional 6 months. Tumor recurrence will be evaluated up to 3 years after training initiation.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients diagnosed with liver metastasis and scheduled for liver metastasis surgical resection

Exclusion Criteria:

* Age <18
* Pregnancy
* Physical or mental disabilities that prohibit execution of test or training procedures
* Inability to understand the Danish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen consumption (VO2peak) | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in VO2peak assessed during an incremental exercise test to volitional exhaustion on a bicycle ergometer

SECONDARY OUTCOMES:
3-years recurrence-free survival | Randomization to 3 years after randomization
  Proportion of patients who survive without relapse (formation of new tumors) for the 3-year period
3-years overall survival | Randomization to 3 years after randomization
  Proportion of patients who are alive 3 years after randomization
Changes in Aerobic Capacity: Ventilatory threshold | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in ventilatory threshold assessed during an incremental exercise test to volitional exhaustion on a bicycle ergometer
Changes in Aerobic Capacity: Peak power output | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in peak power output assessed during an incremental exercise test to volitional exhaustion on a bicycle ergometer
Changes in Muscle strength: Hand grip strength | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in hand grip strength, assessed using a dynamometer
Changes in Muscle strength: Leg press maximal muscle strength | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in leg press one repetition maximum (1RM)
Changes in Functional performance: Habitual gait speed | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in habitual gait speed
Changes in Functional performance: Maximal gait speed | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in maximal gait speed
Changes in Functional performance: Stair climbing performance | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in time required to climb a specific staircase
Changes in Functional performance: 30 seconds Sit-to-stand | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in the number of stands from sitting position that can be performed during 30 seconds
Changes in Body composition and anthropometrics: Body mass | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in body mass
Changes in Body composition and anthropometrics: Total lean mass | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in total lean mass assessed by dual energy x-ray absorptiometry (DXA)
Changes in Body composition and anthropometrics: Total fat mass | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in total fat mass assessed by DXA
Changes in Body composition and anthropometrics: Bone mineral density | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in bone mineral density assessed by DXA
Changes in Body composition and anthropometrics: Waist circumference | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in waist circumference
Changes in Body composition and anthropometrics: Hip circumference | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in Hip circumference
Changes in Systolic Blood pressure | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting systolic blood pressure
Changes in Diastolic Blood pressure | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting diastolic blood pressure
Changes in Heart rate | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting heart rate
Changes in Blood biochemistry: leukocyte differential counts | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting leukocyte differential counts (total and per type [eosinophils, basophils, lymphocytes, monocytes, neutrophils])
Changes in Blood biochemistry: C-reactive protein | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting C-reactive protein levels in blood
Changes in Blood biochemistry: Insulin | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting insulin blood levels
Changes in Blood biochemistry: Glucose | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting glucose blood levels
Changes in Blood biochemistry: Triglycerides | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting triglycerides blood levels
Changes in Blood biochemistry: LDL-Cholesterol | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting LDL-cholesterol blood levels
Changes in Blood biochemistry: HDL-Cholesterol | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting HDL-cholesterol blood levels
Changes in Cytokine levels in blood: Interleukin-6 | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting Interleukin-6 blood levels
Changes in Cytokine levels in blood: Interleukin-1 | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting Interleukin-1 blood levels
Changes in Cytokine levels in blood: Interleukin-7 | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting Interleukin-7 blood levels
Changes in Cytokine levels in blood: Interleukin-8 | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting Interleukin-8 blood levels
Changes in Cytokine levels in blood: Interleukin-15 | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting Interleukin-15 blood levels
Changes in Cytokine levels in blood: Interleukin-1β | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting Interleukin-1β blood levels
Changes in Cytokine levels in blood: Interleukin-10 | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting Interleukin-10 blood levels
Changes in Cytokine levels in blood: Tumor-necrosis-factor alpha (TNFalpha) | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting TNFalpha blood levels
Changes in Cytokine levels in blood: Interferon gamma (IFN-gamma) | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting IFN-gamma blood levels
Changes in Immune cells in blood: Natural killer (NK) cells | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting NK cells
Changes in Immune cells in blood: CD4 T cells | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting CD4 T cells
Changes in Immune cells in blood: CD8 T cells | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting CD8 T cells
Changes in Immune cells in blood: B cells | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting B cells
Changes in Osteonectin | Baseline, 3-, 6-, 9- and 12 months after exercise training initiation
  Changes in resting osteonectin blood levels
Changes in Patient-reported symptomatic adverse events | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Patient-reported symptomatic adverse events, assessed using the using the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Changes in Health-related quality of life: Physical well-being | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported physical well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-28, the higher the score the better quality of life)
Changes in Health-related quality of life: Social well-being | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported social well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-28, the higher the score the better quality of life)
Changes in Health-related quality of life: Emotional well-being | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported emotional well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-24, the higher the score the better quality of life)
Changes in Health-related quality of life: Functional well-being | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported functional well-being assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-28, the higher the score the better quality of life)
Changes in Health-related quality of life: General | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported general health-related qualify of life assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-108, the higher the score the better quality of life)
Changes in Health-related quality of life: Colorectal cancer specific | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported colorectal-cancer specific health-related quality of life assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-28, the higher the score the better quality of life)
Changes in Health-related quality of life: total score | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported in health-related quality of life (total score) assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-136, the higher the score the better quality of life)
Changes in Health-related quality of life: Trial outcome index | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported trial outcome index assessed using the Functional Assessment of Cancer Therapy - Colorectal (FACT-C) (scale scoring 0-84, the higher the score the better quality of life)
Changes in Health-related quality of life: Fatigue | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported fatigue assessed using the Functional Assessment of Cancer Therapy - Fatigue scale (FACIT-Fatigue) (scale score: 0-52, the higher the score the less fatigue)
Changes in Depression | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported depression, assessed using the Hospital Anxiety and Depression Scale (HADS) (scale scoring: 0-21, the higher the score the worse the condition)
Changes in Anxiety | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported anxiety, assessed using the Hospital Anxiety and Depression Scale (HADS) (scale scoring: 0-21, the higher the score the worse the condition)
Changes in Physical activity: Walking | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported weekly duration of walking, assessed using the International Physical Activity Questionnaire (IPAQ)
Changes in Physical activity: Moderate intensity physical activity | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported weekly duration of moderate intensity physical activity, assessed using the International Physical Activity Questionnaire (IPAQ)
Changes in Physical activity: Vigorous intensity physical activity | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported weekly duration of vigorous intensity physical activity, assessed using the International Physical Activity Questionnaire (IPAQ)
Changes in Physical activity: Total intensity physical activity | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported weekly duration of total intensity physical activity, assessed using the International Physical Activity Questionnaire (IPAQ) (Expressed as metabolic equivalent (MET)-min per week: MET level x minutes of activity x events per week)
Changes in Physical activity: sitting time | Baseline, 3-, 6-, 9-, 12-, 24- and 36 months after exercise training initiation
  Changes in patient-reported weekly sitting time, assessed using the International Physical Activity Questionnaire (IPAQ)
Changes in Circulating tumor DNA (ctDNA) | Baseline, 6-, and 12 months after exercise training initiation
  Changes in ctDNA in blood
Changes in DNA methylation | Baseline, 6-, and 12 months after exercise training initiation
  Changes in DNA methylation derived from blood
Changes in treatment tolerance: Relative dose intensity (RDI) of adjuvant chemotherapy | From date of planned initiation to end of adjuvant chemotherapy
  RDI (%) of adjuvant chemotherapy, calculated as the actual dose intensity / standard dose intensity x 100%
Postoperative hospital admissions | From discharge to 12 months after exercise training initiation
  Incidence of postoperative hospital re-admissions, defined as any non-scheduled ≥ 24 h hospitalization
Postoperative complications | From discharge to 30 days after discharge
  Incidence of postoperative complications up to 30 days after surgery (total and by grade and type), assessed using the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Casper Simonsen, PhD, Principal Investigator — Group Leader
Locations (1):
- Rigshospitalet (CFAS), Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No